CLINICAL TRIAL: NCT06761846
Title: A Phase II Study of Sintilimab Combined With Chemotherapy as Postoperative Adjuvant Treatment for Phase III Gastric Adenocarcinoma (GC) and The Adenocarcinoma of Esophagogastric Junction (GEJ)
Brief Title: Sintilimab Combined With Chemotherapy as Adjuvant Treatment for Phase III GC and GEJ
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4947
Record Dates: First submitted 2024-12-28; First posted 2025-01-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-01

CONDITIONS: Gastric Adenocarcinoma; Esophagogastric Junction Adenocarcinoma
MeSH Terms: interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab + SOX/XELOX (Experimental): The study only has one experimental cohort that the subjects who enter the study will receive Sintilimab combined with SOX/XELOX up to 8 cycles, and then receive Sintilimab combined with Tegafur, Gimeracil and Oteracil Potassium Capsules or Capecitabine up to a year ( totally 16 cycles).
  Interventions: Biological: Sintilimab plus Chemotherapy

INTERVENTIONS:
Biological: Sintilimab plus Chemotherapy — chemotherapy includes SOX and XELOX

SUMMARY:
This study is a prospective, single-arm, phase II clinical study. Screening patients with stage III GC/GEJ adenocarcinoma after D2 or broader radical resection. After enrolling in the study, the subjects receive Sintilimab combined with oxaliplatin+Tegafur, Gimeracil and Oteracil Potassium Capsules (SOX) or oxaliplatin+Capecitabine (XELOX) , in which the combined chemotherapy is up to 8 cycles, and the total course of treatment was 16 cycles. The following-up of subjects includes adverse events、disease status、living conditions and the quality of life.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, phase II clinical study. Screening patients with stage III GC/GEJ adenocarcinoma after D2 or broader radical resection that meets the criteria for group entry and does not meet the exclusion criteria. After signing the informed consent, the subjects entered the trial group to receive adjuvant treatment with Sintilimab combined with chemotherapy (SOX or XELOX ), in which SOX or XELOX chemotherapy was up to 8 cycles, and the total course of treatment was 16 cycles. The efficacy is evaluated every 4 cycles during the study treatment. The frequency of follow-up after treatment is defined as: once every 3 months within 2 years after surgery, every 6 months for 2 to 5 years, and once a year after 5 years. The follow-up interval can be adjusted according to the clinical need. Safety follow-up is from the beginning of the first treatment to 30 days after the last medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.
2. Patients with histopathological confirmed gastric/GEJ adenocarcinoma.
3. The pTNM is confirmed between IIIA-IIIC and the PD-L1 CPS>=1.
4. Patients treated with D2 surgery.
5. ECOG is 0 or 1.
6. Patients who could tolerate chemotherapy combined with immunotherapy.
7. Patients who are not pregnant and have no willing to get pregnant within 6 months after the treatment is over.
8. Patients who are willing to offer their postoperative tumor tissue and their peripheral blood samples.
9. Patients who are volunteer to sign the ICF.

Exclusion Criteria:

1. Patients who had received neoadjuvent treatments before surgery.
2. Patients who have discovered tumor relapse or metastasis before adjuvent treatment.
3. Patients who have other malignant tumors.
4. Patients who could not swallow the tablets and capsules.
5. Other conditions which the researchers think are not suitable for participate the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival(DFS) rate | From the time of first dose of adjuvant treatment to the 3 years of the same day
  The disease free survival rate of 3 years after receiving the first dose of treatment

SECONDARY OUTCOMES:
DFS | From the time of first dose of adjuvant treatment to the time when the subjects have confirmed disease progress
  disease free survival
overall survival (OS) | From the time of first dose of adjuvant treatment to the time when the subjects have died for all causes
  overall survival
safety | collect all adverse events since the last medication up to 30 days
  treatment safety and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: LIN YANG, Doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hodpital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No